CLINICAL TRIAL: NCT05960877
Title: The Risk Factors of Thrombosis in Complicated Arteriovenous Fistula in Patients on Regular Hemodialysis
Brief Title: The Risk Factors of Thrombosis in Complicated Arteriovenous Fistula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Aldosouky, Resident doctor, Assiut University
Other Study IDs: AV fistula thrombosis
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arteriovenous Fistula Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
study the risk factors of thrombosis in thrombosed arteriovenous fistula in patients on regular hemodialysis

DETAILED DESCRIPTION:
The number of patients being treated for kidney failure continues to increase every year at a significantly higher rate than that of the world population.

The main renal replacement therapy was hemodialysis (HD) in 57% patients and peritoneal dialysis in 5% patients, while 37% patients underwent a functional kidney transplant.

Native arteriovenous fistula (AVF) is currently the best VA when technically feasible, according to the international dialysis guidelines.

Hemodialysis vascular access failure is the dominant cause of morbidity and the major cost of care for end-stage renal disease (ESRD) patients .

Complications such as thrombosis of VA remain the main problem for many patients with kidney failure.

Since 1994, prospective and case-control studies have explored the relationship between risk factors and arteriovenous fistula thrombus (AVFT) in patients undergoing HD .

Until now, these studies and reviews have revealed that numerous risk factors are associated with AVFT .

Risk factors like arterio-venous graft, age, female sex, C-reactive protein level, fistula site (distal), hypertension and the use of eprex can be associated with AVFT, and this knowledge advances the understanding of AVFT, facilitates multivariable risk prediction profiling, and lays the foundation for future preventive strategies .

ELIGIBILITY:
Inclusion Criteria:

* All patients on maintenance hemodialysis treatment at the dialysis unit of the department of nephrology in Assiut University Hospital .

Exclusion Criteria:

* Patients with known other risk factors of thrombosis, e.g., malignancy, pregnancy, cocs and nephrotic syndrome.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients on maintenance hemodialysis treatment at the dialysis unit of the department of nephrology in Assiut University Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of the risk factors of thrombosis in complicated AV Fistula in patients on regular hemodialysis | 1 week following AV Fistula occlusion
  Provide the evidence on the association between potential risk factors and arteriovenous fistula thrombus

REFERENCES:
- [Background] Zhang Y, Yi J, Zhang R, Peng Y, Dong J, Sha L. Risk Factors for Arteriovenous Fistula Thrombus Development: A Systematic Review and Meta-Analysis. Kidney Blood Press Res. 2022;47(11):643-653. doi: 10.1159/000526768. Epub 2022 Sep 16. PMID 36116428
- [Background] Goldwasser P, Avram MM, Collier JT, Michel MA, Gusik SA, Mittman N. Correlates of vascular access occlusion in hemodialysis. Am J Kidney Dis. 1994 Nov;24(5):785-94. doi: 10.1016/s0272-6386(12)80672-x. PMID 7977320
- [Background] Fila B. Quality indicators of vascular access procedures for hemodialysis. Int Urol Nephrol. 2021 Mar;53(3):497-504. doi: 10.1007/s11255-020-02609-5. Epub 2020 Aug 31. PMID 32869172
- [Background] Fekih-Mrissa N, Sayeh A, Baffoun A, Beji M, Mrad M, Hmida J, Nsiri B. Association Between Thrombophilic Gene Mutations and the Risk of Vascular Access Thrombosis in Hemodialysis Patients. Ther Apher Dial. 2016 Apr;20(2):107-11. doi: 10.1111/1744-9987.12379. Epub 2016 Mar 23. PMID 27004938
- [Background] Vascular Access 2006 Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S176-247. doi: 10.1053/j.ajkd.2006.04.029. No abstract available. PMID 16813989
- [Background] Feldman HI, Kobrin S, Wasserstein A. Hemodialysis vascular access morbidity. J Am Soc Nephrol. 1996 Apr;7(4):523-35. doi: 10.1681/ASN.V74523. PMID 8724885
- [Background] Salahi H, Fazelzadeh A, Mehdizadeh A, Razmkon A, Malek-Hosseini SA. Complications of arteriovenous fistula in dialysis patients. Transplant Proc. 2006 Jun;38(5):1261-4. doi: 10.1016/j.transproceed.2006.02.066. PMID 16797276